CLINICAL TRIAL: NCT05874362
Title: People Bereaved by Violent Death : a Negative Event Biases and Temporal Perception Study
Brief Title: People Bereaved by Violent Death : Negative Event Biases and Temporal Perception
Acronym: PrEVENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2023-A00304-41
Record Dates: First submitted 2023-05-12; First posted 2023-05-24 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Subjects will be separated into two groups at the end of the study to conduct analyses, depending on the development of a psychiatric complication or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with complications at 3 month (Other): Group composed with participants who develop a psychiatric complication (depressive episode or post traumatic stress disorder) 3 month after the death of their loved one.
  Interventions: Other: Diagnosis of depressive episode or post traumatic stress disorder
- Group without complication at 3 month (Other): Group composed with participants who do not develop a psychiatric complication (depressive episode or post traumatic stress disorder) 3 month after the death of their loved one.
  Interventions: Other: No diagnosis of depressive episode or post traumatic stress disorder

INTERVENTIONS:
Other: Diagnosis of depressive episode or post traumatic stress disorder — Clinical diagnosis of depressive episode or post traumatic stress disorder, confirmed
  Arms: Group with complications at 3 month
Other: No diagnosis of depressive episode or post traumatic stress disorder — No elements in clinical assessment for the diagnosis of a depressive episode or post traumatic stress disorder
  Arms: Group without complication at 3 month

SUMMARY:
A violent death is defined by its brutality, unexpectedness and is secondary to an external cause (suicide, homicide, accident). Bereavement following a violent death constitutes a particular clinical situation, at risk of complications. Research on bereavement after a violent death shows higher risks of psychiatric and somatic complications than in bereavement by non-violent death. These complications, sometimes comorbid, take the form of depressive episodes, post-traumatic stress disorders, suicidal behavior and prolonged grief disorders after 12 months, precociously mediated by ruminations.

Processes responsible for this increased risk of complications are poorly documented. Current literature relates mainly to socio-demographic and epidemiological factors which, alone, do not explain this difference in risks. Further research is needed exploring other kinds of data and processes. To our knowledge, there is no description of early neurocognitive functioning in people bereaved after violent death. This study aims at exploring early neurocognitive processes which can lead to complications in people bereaved by violent death.

DETAILED DESCRIPTION:
This work is based on cognitive models of post-traumatic stress disorder involving cognitive biases as factors of development and maintenance of symptomatology. Indeed, in people exposed to a potentially traumatic event, it has been found that an early deterioration in cognitive functioning is a risk factor for developing post-traumatic stress disorders . Among these cognitive alterations, attentional biases toward threat are the most explored and research shows both facilitated engagement and difficulties in disengagement in front of threatening stimuli. In addition, while expecting for a negative event, there is changes in the perception of time . These processes can be explored on a behavioral level and in electroencephalography , in particular through the evoked related potentials following a stimulus. Among these evoked related potentials , the Late Positive Potential component reflects the attentional process, while the Contingent Negative Variation component and the α and β power reflects temporal perception.

As exposure to violent death can have a traumatic impact, our hypothesis is that people bereaved by violent death could present attentional biases, and that these biases would be prodromal of the onset of a psychiatric disorder (Post-traumatic stress disorders , depression afterwards). The objective of this study is to describe the presence of these biases through electrophysiological and behavioral measures in a sample of subjects bereaved by violent death.

ELIGIBILITY:
Inclusion Criteria:

* An age between 18 and 65 years old
* Recent bereavement by violent death of a relative in first and second degree

Exclusion Criteria:

* Protected adults
* Lack of mastering French language
* History of neurodegenerative disorder
* History of psychiatric disorder treated pharmacologically with modification of the basic treatment in the month preceding the death
* The take of an benzodiazepine treatment in the 24th hours before the first visit (T0)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Amplitude of the Late Positive Potential (LPP) component in unpredictable event condition | Between Day15 and Day30 after the death of one's loved one
  Measure in Electroencephalography (EEG) of the Late Positive Potential (LPP), an Event Related Potential (ERP) relating to attention biases

SECONDARY OUTCOMES:
Amplitude of the Contingent Negative Variation (CNV ) component in unpredictable event condition | Between Day15 and Day30 after the death of one's loved one
  Measure in Electroencephalography (EEG) of the Contingent Negative Variation (CNV), EEG measures relating to temporal perception
Amplitude of the alpha and beta power in unpredictable event condition | Between Day15 and Day30 after the death of one's loved one
  Measure in Electroencephalography (EEG) of the alpha and beta power, EEG measures relating to temporal perception
Comparison of Constant Errors (CE) relative to time estimates in the unpredictability condition (D15-J30) in people developing a psychiatric complication at 3 months and in people not developing these complications. | Between Day15 and Day30 after the death of one's loved one
  Proportion of overestimation of the duration preceding an unpredictable event, and calculation of the point of subjective equality, for measurements of constant errors (CEs) corresponding to the difference between the effective time and the point of subjective equality for each subject

CONTACTS AND LOCATIONS:
Overall Officials: Edouard LEAUNE, Principal Investigator — Vinatier Hospital
Locations (1):
- Hopital Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: No